CLINICAL TRIAL: NCT04366401
Title: Efficacy of Dietary Modulation With High Prebiotic and Probiotic Content on Nutritional and Metabolic Status in Schizophrenia Spectrum Disorders
Brief Title: Efficacy of Prebiotic and Probiotic Dietary Modulation in Schizophrenic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Principal Investigator, Alfonso Sevillano Jiménez, Registered Nurse, Psychiatric-Mental Health Nurse Practitioner, Master Of Science, Doctoral Student, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UC-Psychobiotics2020
Record Dates: First submitted 2020-04-18; First posted 2020-04-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia and Related Disorders; Diet Habit
Keywords: Prebiotic; Probiotic; Schizophrenia Spectrum and Other Psychotic Disorders; Diet Therapy
MeSH Terms: conditions — Schizophrenia; Feeding Behavior; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Two-arm, double-blind, randomized clinical trial in balanced blocks of six months of intervention will be developed in a group of 50 individuals (25 for the intervention group -IG-,25 for the control group -CG-). The GC will receive conventional dietary advice on an individual basis. In the IG, an individual diet-nutrition education program with high prebiotic and probiotic content will be established. Data on psychopathological status (PANSS and PSP scales), and blood tests (haemogram, lipid profile, etc.),at the beginning, after three and six months. The estimate of intestinal microbiota and the usual nutritional pattern will be assessed at baseline and at six months, using a stool test and a validated food frequency questionnaire, respectively. To assess the degree of adherence, IG participants will fill in a specific weekly record of the main dishes/foods consumed. Anthropometric parameters will be analysed monthly (BMI, blood pressure, heart rate, abdominal perimeter).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Dietary Advice (Active Comparator): The control group will consist of participants diagnosed on the schizophrenic spectrum who will receive conventional dietary counseling (n=25) on an individual basis.
  In the control group, data will be collected on the psychopathological state (PANSS and PSP scales), and blood analysis (hemogram, lipid profile, etc.). The measurements will be taken at the beginning (basal), at three and six months. The estimation of the intestinal microbiota and the usual nutritional pattern will also be evaluated at the beginning and at six months, using a stool test and a validated food frequency questionnaire, respectively. To assess the degree of adherence, GI participants will fill in a specific weekly record of the main dishes/foods consumed. At least, anthropometric parameters will also be analysed monthly (BMI, blood pressure, heart rate, abdominal perimeter).
  Interventions: Behavioral: Conventional Dietary Advice
- Prebiotic/Probiotic Dietary Modulation (Experimental): In the intervention group (n=25), individual dietary counseling will be established through intensive nutritional counseling to provide a high prebiotic and probiotic food pattern.
  In the experimental group, data will be collected on psychopathological status (Positive and Negative Syndrome Scale -PANSS- and Personal and Social Functioning Scale -PSP-), and blood tests (haemogram, lipid profile, etc.). The measurements will be taken at the beginning (basal), at three and six months. The estimation of the intestinal microbiota and the usual nutritional pattern will also be evaluated at the beginning and at six months, using a stool test and a validated food frequency questionnaire, respectively. To assess the degree of adherence, GI participants will fill in a specific weekly record of the main dishes/foods consumed. At least, anthropometric parameters will also be analysed monthly (BMI, blood pressure, heart rate, abdominal perimeter).
  Interventions: Behavioral: Prebiotic/Probiotic Dietary Modulation

INTERVENTIONS:
Behavioral: Conventional Dietary Advice — The education content in the control group will be centered on the acquisition of knowledge about:
  * - Underlying mental pathology, lifestyles and associated comorbidities
  * - Immediate principles: Carbohydrates, lipids, proteins, fiber, vitamins, and minerals; energy needs; consumption requirements.
  * - Water requirements.
  * - Foodstuffs.
  * - Culinary techniques: conservation of properties of the diet.
  * - Feeding in particular situations.
  Arms: Conventional Dietary Advice
Behavioral: Prebiotic/Probiotic Dietary Modulation — The education content in the intervention group will be based on general principles of conventional dietary advice in an intensified manner, centered on the acquisition of specific knowledge about:
  * - Underlying mental pathology, lifestyles and associated comorbidities
  * - Immediate principles: Carbohydrates, lipids, proteins, fiber, vitamins, and minerals; energy needs; consumption requirements.
  * - Water requirements.
  * - Foodstuffs.
  * - Description and justification of prescribed prebiotic and probiotic diet.
  * - Culinary techniques: conservation of properties of the prebiotic and probiotic diet.
  * - Optimal distribution and interchange of foods with high prebiotic and probiotic content.
  * - Feeding in particular situations.
  Arms: Prebiotic/Probiotic Dietary Modulation

SUMMARY:
The microbiota plays a vital role in the two-way communication between the gastrointestinal tract and the central nervous system (CNS), articulated as the microbiota-intestine-brain axis. This function provides sufficient evidence to establish a causal relationship between numerous neuropsychiatric disorders, such as schizophrenia. Besides, the microbiota modulation through the dietary pattern is related to the improvement of the physical and psychopathological health of patients. In this sense, the use of psychobiotics (prebiotics and probiotics with nutraceutical action) highlights. This research will be aimed to test the efficacy of prebiotic dietary modulation in patients diagnosed with schizophrenia, attending to the impact in nutritional and cardio-metabolic conditions. In this sense, two-arms, double-blind, randomized in balanced blocks clinical trial of six months of intervention, will be developed in a group of 50 individuals (25 for the intervention group (IG) and 25 for the control group). First, an initial group session will be held to present the purpose of the research, as well as each of the relevant aspects during its development. Similarly, certain focus groups will be established periodically to redefine and guide the improvement of the development of the investigation, ensuring adequate compliance with the study after the implementation of the diet and nutrition education program. The dietary education will be designed and supervised by qualified personnel with recognized competencies for this type of intervention (nurses and dietitians). The CG will be made up of those participants who receive conventional dietary advice individually in serial consultations. On the other hand, in the IG, this intervention will be characterized by the establishment of an individual program of dietetic-nutritional education with high prebiotic and probiotic content. During the development of the study, data will be collected on the psychopathological state (PANSS and PSP scales), and blood test (hemogram, lipid profile, etc.). Measures will be taken at the beginning (basal), at three and six months. The estimation of intestinal microbiota and the usual nutritional pattern will also be assessed at the beginning and six months, using a stool test and a validated Food Frequency Questionnaire (FFQ), respectively. To evaluate the degree of adherence, participants in the IG will fill a specific weekly record of the main dishes/food consumed. At least, anthropometric parameters will also be analyzed monthly (BMI, blood pressure, heart rate, abdominal perimeter).

DETAILED DESCRIPTION:
1. INTRODUCTION

   1.1. Theoretical Framework

   Schizophrenia is a chronic mental illness characterized by significant clinical heterogeneity and a long evolution over time, determined by periods of psychotic exacerbation and phases of stabilization. The semiology of this nosological entity is established in positive and negative symptoms, with variable levels of dysfunction and clinical presentation, and having an essential impact on the patient's quality of life. Similarly, surrounding the schizophrenic spectrum, the existence of the associated neurocognitive impairment stands out, prevailing the disorders of social and occupational functioning, as well as a significant degree of disorganization.

   Many theories have tried to elucidate the origin of schizophrenia, where the complexity of its etiopathogenesis is a determining factor in establishing an appropriate, specific, and effective therapeutic approach. However, despite numerous defined aetiological premises, the dopaminergic hypothesis is considered the final common pathway of all of them, converging numerous associated pathogenic mechanisms, where low-grade systemic inflammation and oxidative stress stand out.

   Undoubtedly, the traditional therapeutic approach has perceived the role of nutrition as a minor intervention in psychiatry, especially in psychotic disorders such as schizophrenia. However, the advances established in the last decade, mainly associated with the development of the holobionte theory and the evolution of metagenomics, as well as the presence of new dietary patterns of low nutritional quality in different western societies, have contributed significantly to the global understanding of the role of nutritional patterns on the functioning of the Central Nervous System (CNS), as well as on the possible mechanisms or etiological pathways of psychiatric disorders.

   In this regard, it is necessary to highlight the role of the intestinal microbiota (IM) and the intimate relationship it exerts on the numerous functions of the body, such as the development and maturation of the CNS, nutrition, immune response or systemic inflammation. This effect is carried out through various established communication pathways: vagal nerve (primary), intestinal hormones, cytokines, exosomes, and microRNAs. Thus, the existence of possible modifications in the concentration of this biota (considering average concentrations around 10^13 CFU/g), may trigger homeostatic alterations or aggravate pathogenic conditions, a fact commonly called dysbiosis. This concentration of microbiota is fundamentally determined by dietary patterns, genetic factors, iatrogenic antibiotherapy, type of breastfeeding (maternal or formula), age, exercise, and continuous stress, among others.

   As a consequence of these discoveries, the concept of the "Microbiota-Intestine-Brain Axis" emerges. This term refers to the two-way communication pathway established between the CNS, the gastrointestinal tract, and the MI, mediated by the microbial metabolites of dietary products such as dietary fiber, tryptophan or arginine, as well as by endocrine and neuronal mechanisms. The close relationship established between MI and the CNS lies in the production of a multitude of neurotransmitters essential for normal neuronal functioning, such as serotonin, GABA, dopamine or noradrenaline, among others. Similarly, MI exerts essential trophic, metabolic, and protective functions, which are a determining factor in the normal neuropsychiatric function.

   Thus, according to the theory of low-grade systemic inflammation, when a state of dysbiosis occurs in the symbiote MI, it generates a cascade of pro-inflammatory agents, such as lipopolysaccharide (LPS), a bacterial endotoxin, capable of modifying both the integrity and the permeability of enterocytes. This alteration triggers the release of pro-inflammatory cytokines (tumor necrosis factor ἀ [TNF-ἀ] or interleukins type 6 or 1ß [IL-6, IL-1ß], both capable of altering intestinal tissue integrity), originating synergies between inflammation, increased oxidative stress and imbalance of energetic homeostasis. This cascade of reactions causes an increase in neurodegeneration and excitotoxicity, mediated by the vagus nerve. Thus, it has been shown that the activation of a state of low inflammation is related to a worse prognosis of schizophrenia concerning positive and negative symptoms, cognitive performance, and loss of brain volume. Similarly, alterations in specific pro-inflammatory cytokines or state markers have been described, especially in psychotic relapses or prodromal phases (IL-6, TGF-ß, among others), as well as a decrease in their concentration after the introduction of antipsychotic treatment, with consequent clinical improvement.

   1.2. Justification

   Existing scientific production shows a high rate of disability and morbimortality in people suffering from some psychiatric disorder concerning the rest of the general clinical population, especially in those patients with a severe and long-term mental disorder (LTMD), highlighting dysfunctions of the psychotic and affective spectrum: schizophrenia and bipolar disorder (respectively). This morbidity and mortality rate in the psychiatric population is up to 20% higher and, quantitatively, represents an average of 25 years of life lost. Besides, patients with LTMD have a life expectancy of less than 20% (57 years in men and 65 years in women). It is estimated that the relative risk (RR) of this disease is 2.41 higher for mortality from any causes, these being mainly comprised of cardiovascular, infectious, respiratory, and endocrine diseases (60% of premature deaths in this clinical population). Also, the leading established causes of mortality are closely linked to the development of the Metabolic Syndrome (MS), also called insulin resistance syndrome. The MS is considered a determining factor in the physical health of the patient, tripling the incidence of cardio-metabolic diseases.

   The main etiopathogenic determinants of this fact are the factors inherent to the disease itself, as well as genetic factors, resistance to adequate care in terms of physical health and lifestyles followed by these patients (far removed from those considered healthy).

   Despite the magnitude and severity of the problem, interventions aimed to modify lifestyles do not play an essential role in therapy and are not part of the usual clinical practice with the psychiatric population. This fact could be explained by the lack of understanding of the multiple mechanisms and etiological factors involved in the neurogenesis of schizophrenia, and leads to a multidisciplinary approach, but essentially psychopharmacological and psychotherapeutic. It is, therefore, vital to address modifiable factors such as dietary patterns, which have evidenced to be an efficient therapeutic intervention to improve both the psychopathological dysfunction and the physical health of the subjects and can be considered as an addition to the conventional therapeutic approach.

   In this sense, some dietary interventions carried out to modulate intestinal microbiota in psychotic disorders through the use of so-called "psychobiotics". This term refers to the set of substances that include probiotics and/or prebiotics and whose administration causes health benefits in psychiatric patients. Probiotics include microorganisms of the intestinal biota, which, provided in adequate quantities, offer a benefit for the host (highlighting the genera Lactobacillus and Bifidobacterium, among others). On the other hand, prebiotics are non-digestible dietary fiber (mainly fructooligosaccharides and oligosaccharides, inulin or pectins), which are substances that promote optimal growth and development of probiotics in the gastrointestinal tract, reducing pathogenic microbiota, through the production of short-chain fatty acids (SCFA).

   It is worth noting the growing effort to highlight the role played by prebiotics and or probiotics in the microbiota-intestine-brain axis, which is currently a relevant object of study. In this regard, adequate dietary planning in psychiatric patients with psychopathological dysfunction and at risk of iatrogenic metabolic syndrome, could be considered as a therapy of choice in these subjects, improving altered clinical patterns and difficulties in the patient's vital and functional performance. Similarly, adequate nutritional management could be used as an adjunct to antipsychotic pharmacotherapy and the cardio-metabolic approach, reducing the number of homeostatic drugs or even replacing them in cases of intolerance in the target population.

   In short, the future of the development of Mental Health is determined by the need for a multimodal approach, where nutritional factors represent the cornerstone in achieving optimal results in health, level of functionality, and, therefore, quality of life of patients. Likewise, dietary modulation has the added value of improving the morbidity and mortality associated with schizophrenia, with optimal levels in terms of cost-effectiveness, better than those shown by the approaches currently used.
2. RESEARCH QUESTION AND OBJECTIVES

   Could the modulation of the dietary pattern through the optimal incorporation of prebiotics and probiotics improve the nutritional and cardio-metabolic status of patients diagnosed with schizophrenia spectrum disorders, as well as improve their clinical impact in psychopathological terms?

   2.1. Research hypotheses or assumptions

   The integration of non-digestible dietary fiber and fermented dairy products into the conventional eating pattern of the psychiatric population diagnosed with schizophrenia (in any of its variants), can improve the nutritional status and, consequently, the level of physical health of these patients. Likewise, this prebiotic and probiotic content would allow the improvement of the psychopathological state in those clinical areas altered by the underlying mental disorder.

   2.2. Objectives

   2.2.1. Main objective

   - Determination of the nutritional and cardio-metabolic efficacy of a prebiotic and probiotic dietary intervention in patients with schizophrenia spectrum disorders

   2.2.2. Specific objectives
   * To determine the baseline nutritional status of the target population.
   * To identify the usual dietary patterns in this population, clarifying the nutritional value of the main dishes consumed, as well as their link with the physical health status of individuals.
   * To know the existing scientific evidence regarding the construction of determinants (explicit and implicit) that influence the microbiota-intestine-brain axis.
   * To evaluate the psychopathological impact of the incorporation of prebiotics and probiotics in the habitual dietetic-nutritional pattern in patients diagnosed with the spectrum of schizophrenia.
   * To evaluate the cardio-metabolic impact of a standardized dietary planning with high prebiotic and probiotic content, adapted to the inherent characteristics of the psychiatric population.
   * To develop and validate a program that allows for the detection of areas of improvement, establishing assessment strategies, and an appropriate action plan in Mental Health, which allows for adequate dietary care through the use of psychobiotics.
3. MATERIAL AND METHODS

   3.1. Study design

   A two-arms, double-blind, randomized in balanced blocks clinical trial of six months of intervention, will be carried out in psychiatric patients diagnosed with schizophrenic spectrum disorders (without distinction by type) -n=50-. The control group will be made up of those participants who will receive conventional dietary advice (n=25) on an individual basis. In the intervention group (n=25), this advice will be established individually through intensive nutritional guidance offering a food pattern with a high prebiotic and probiotic content. In both intervention groups, educational material of visual support will be used during the sessions. The dietary intervention will be designed and supervised by qualified personnel with recognized competencies for this type of intervention (nurses and dietitians) and will be agreed upon through serial interviews and focus groups. In this sense, these focus groups will be applied to improve the established dietetic-nutritional intervention, guaranteeing its correct adaptation, according to the study population.

   The study will begin with a group session for the presentation of the research project in the health center and/or psychiatric service consultation. During the development of the study, data will be collected on the psychopathological state (Positive and Negative Syndrome Scale -PANSS- and Personal and Social Functioning Scale -PSP- scales), and blood test (hemogram, lipid profile, etc.). Measures will be taken at the beginning (basal), at three and six months. The estimation of intestinal microbiota and the usual nutritional pattern will also be assessed at the beginning and six months, using a stool test and a validated Food Frequency Questionnaire (FFQ), respectively. To evaluate the degree of adherence, participants in the IG will fill a specific weekly record of the main dishes/food consumed. At least, anthropometric parameters will also be analyzed monthly (BMI, blood pressure, heart rate, abdominal perimeter).

   3.2. Statistical analysis

   Quantitative variables will be presented with mean and standard deviation, and qualitative variables will be shown in frequencies and percentages.

   The Kolmogorov-Smirnov test will be used to compare the goodness of fit to a normal distribution of data from quantitative variables. For the contrast of bivariate hypotheses, the Student t-test will be performed for two means, while for qualitative variables, the Chi-Square and Fisher's exact test will be used, when necessary. Likewise, for the analysis of three or more means, the ANOVA of repeated means will be used. On the other hand, the correlation between quantitative variables will be verified through the Pearson's coefficient r. Finally, if the criterion of normality or homocedasticity is not met, the non-parametric versions of the above tests shall be performed.

   Logistic regressions will be carried out to determine which variables can determine the improvement of the nutritional pattern and physical health through the Food Frequency Questionnaire, as well as blood and stool analytical values. Similarly, this analysis will be established concerning the psychopathological status through the PSP and PANSS scales, both of which have a discrete quantitative and nominal result values, according to established cut-off points and clinical interpretation. Raw and adjusted odds ratios (ORs) will be calculated. Log-likelihood, the goodness of fit statistic, Cox and Snell R2, Nagelkerke R2, and Hosmer-Lemeshow tests should be used to assess the overall model fit. The exponentiation will be used to calculate the beta coefficients.

   For all statistical analyses, an alpha error probability of less than 5% (p<0.05) will be accepted, and the confidence interval will be calculated at 95%. The software SPSS (version 25.0) and EPIDAT (version 4.2) shall be used for the statistical analysis.
4. WORK PLAN

   An intervention schedule has been established, with a total duration of 6 months, which is divided into three blocks:

   4.1. Block 1

   This first block focuses on the selection of the target population according to inclusion criteria. Firstly, a group session to present the program and the methodology of the study will be carried out. During the first fifteen days of the study, a focus group with professionals to reach a consensus on the intervention will be held. Subsequently, the appropriate modifications will be made to improve and adapt to the dietary and nutritional intervention.

   Consequently, the recruitment and initial psychopathological and nutritional assessment of the participants will be carried out, using the Scale of Positive and Negative Syndromes (PANSS) and the Scale of Personal and Social Functioning (PSP). For the nutritional evaluation, the analytical and anthropometric basal determination of the participating patients will be carried out, as well as the evaluation of the habitual dietary pattern through a validated FFQ and weekly record of the main dishes and foods consumed. Similarly, an estimate of the intestinal bacterial flora is required employing stool culture.

   4.2. Block 2

   The second block includes the implementation of the 6-month individual nutrition education program (associated with two months of educational reinforcement, according to block 3). It will consist of eight sessions, the first four being biweekly, followed by four monthly, to which four sessions of educational reinforcement will be added to the 3 and 5 months of study. The minimum duration of each session has been established for 30 minutes. However, this length could be different, considering the characteristics of the participants. The control group will be made up of those participants who will receive standardized dietary advice. In this sense, the education content in the intervention group will be based on general principles of conventional dietary advice in an intensified manner, centered on the acquisition of specific knowledge about:
   * - Underlying mental pathology, lifestyles and associated comorbidities
   * - Immediate principles: Carbohydrates, lipids, proteins, fiber, vitamins, and minerals; energy needs; consumption requirements.
   * - Water requirements.
   * - Foodstuffs.
   * - Description and justification of prescribed prebiotic and probiotic diet.
   * - Culinary techniques: conservation of properties of the prebiotic and probiotic diet.
   * - Optimal distribution and interchange of foods with high prebiotic and probiotic content.
   * - Feeding in particular situations.

   In both the IG and the CG, visual support resources will be used during the development of the established sessions.

   4.3. Block 3

   Finally, to evaluate the effectiveness of the intervention, the modification in the nutritional, the cardio-metabolic, and the psychopathological area will be assessed. For doing this, researchers will carry out anthropometric determination, clinical evaluation, the performance of stool culture, and the study of the dietary pattern, as the investigators commented above.

   Likewise, in this block, an educational reinforcement (both in IG and CG) of what was treated in Block 2 will be offered, three and five months after the beginning of the block, every 15 days for the IG and monthly for the CG.

   Once the intervention is concluded, the analysis of the collected data will be performed, culminating in the development of the scientific production and the writing of the research report.
5. RESULTS

   5.1.Expected results and outputs

   Firstly, it is expected to obtain the necessary information for the determination of the optimal dietary pattern for those participants in the study, thus allowing the development of a nutritional intervention with high prebiotic and probiotic content, appropriate for the population under study.

   Likewise, the aim is to ensure that all participants improve their health status through the adaptation of the feeding pattern, developing adherence to healthier lifestyles adapted to the conditions of each patient.

   Finally, it is expected to demonstrate that an adequate dietary modulation with a high prebiotic and probiotic content, leads to a significant improvement in the nutritional status and, therefore, the cardio-metabolic, of the participants, mediated by the microbiota-intestine-brain axis. Furthermore, it is presumed to reach a degree of evidence that allows establishing nutritional management as an effective therapeutic intervention in the psychopathological treatment of patients with schizophrenia spectrum disorders, in any of its variants.
6. ETHICAL AND LEGAL IMPLICATIONS

6.1. Risk-benefit analysis

A priori, since the intervention will be based on expert opinion and founded on a solid scientific basis, it is not considered that the participants in this study could be exposed to any risk or discomfort, except the routine health monitoring and control. In this sense, it should be noted that most of the controls established are determined by non-invasive tests (validated questionnaires and scales, anthropometric measurements, stool culture, etc.), minimizing the discomfort caused during the development of the intervention. On the other hand, as an invasive measure, the possible side effects derived from blood extraction by venous puncture should be highlighted. Such effects are established infrequently, but should they appear, including dizziness, pain, or hematomas, among others.

In terms of benefit, regardless of whether participants are assigned to the IG or the CG, the type of intervention carried out, whether it is conventional dietary advice or an educational program with a high prebiotic and probiotic content, will seek to modify lifestyles towards healthier ones, mediated by the improvement of the dietary pattern.

Besides, if it is evident that the participants assigned to the IG present significant results in nutritional, cardio-metabolic and psychopathological terms, a cost-efficient solution will have been found for the health system, allowing people diagnosed with schizophrenic spectrum disorders to have access to lifestyle improvement plans and better tolerability to psychopharmacological treatment. This finding could alleviate the number of psychiatric consultations required by the need for dosage adjustments and/or associated physical health problems. In this way, a solution will be offered to the problems of accessibility (geographical, economic, etc.), level of dysfunctionality and morbimortality, of high incidence in this psychiatric population.

6.2. Ethical principles

The study will be carried out respecting the fundamental principles established in the Declaration of Helsinki (1964), the Council of Europe Convention on Human Rights and Biomedicine (1997), the UNESCO Universal Declaration on the Human Genome and Human Rights (1997). Researches will also follow the requirements established by Spanish legislation (Organic Law 3/2018 of 5 December on the Protection of Personal Data and the Guarantee of Digital Rights and Law 41/2002 of 14 November), which is the fundamental law regulating patient autonomy and rights and obligations in the field of clinical information and documentation. All the information analysed by the principal investigator of this study is subject to the maintenance of professional secrecy.

In any case, each participant will be assigned a code as a registry, where all the relative data will be mechanized in an anonymous way, delimiting the access to the database only to the personnel linked to the development of the study, previous authorization of the investigator in charge of it.

6.3. Informed consent Data will only be collected from those subjects who have previously signed the informed consent form, which is included in the Patient/Legal Representative Information Sheet (ANNEXES: Annex I and II), included in the presentation of the research project.

ELIGIBILITY:
Inclusion Criteria:

* -Patients diagnosed on the spectrum of schizophrenia (without distinction by type), according to criteria DSM-5 and/or ICD-11.
* Age between 18-65 years.
* - Absence of gastrointestinal comorbidity that contraindicates the use of prebiotics and/or probiotics (intolerance, explosive diarrhea, acute abdominal pain, etc.).
* -To show clinical stability for six months before the start of the study (absence of psychiatric hospitalization, maintenance of the level of functionality, and lack of social and occupational absenteeism).
* - To manifest agreement to participate in the study and to sign of informed consent.

Exclusion Criteria:

* -Non-compliance with the inclusion criteria mentioned above.
* - To suffer from somatic or neurocognitive situation that prevents participation and collaboration in the fulfillment of the protocol.
* - To follow standardized dietary planning not modulated by the population under study (catering, institutional or collective feeding, etc.).
* -Concomitant administration of antibiotherapy.
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Changes in Clinical Efficacy of Prebiotic/Probiotic Dietary Modulation in 6 Months of Intervention | Basal, three and six months respectively
  -- Personal and Social Functioning Scale (categorized PSP) outcome: discrete. Scoring interval (range 10 points: 0-100) in relation to the degree of dysfunction of the areas: self-care, personal and social relationships, socially functional activities (work/study), disturbing and aggressive behaviour. To establish the final decimal point of this interval, 10 functional aspects must be scored (YES: 1 point, NO: 0 points). Finally, the higher the score, the better the patient's functional level.
Changes in Clinical Efficacy of Prebiotic/Probiotic Dietary Modulation in 6 Months of Intervention | Basal, three and six months respectively
  -- Scale for Positive and Negative Schizophrenia Syndrome (categorized PANSS): discrete. It provides four dimensional scores: Positive syndrome, Negative syndrome, Compound scale, General psychopathology.
  The score on the positive (PANSS-P) is obtained by adding up the scores of each item. The scores will therefore range from 7 to 49 for the positive scale..
  There are no cut-off points for the direct scores obtained, but these are transformed by means of a conversion table into percentiles. Futhermore, PANSS also provides categorical information, indicating whether the schizophrenic disorder is positive, negative or mixed.
Changes in Clinical Efficacy of Prebiotic/Probiotic Dietary Modulation in 6 Months of Intervention | Basal, three and six months respectively
  -- Scale for Positive and Negative Schizophrenia Syndrome (categorized PANSS): discrete. It provides four dimensional scores: Positive syndrome, Negative syndrome, Compound scale, General psychopathology.
  The score on the negative (PANSS-N) is obtained by adding up the scores of each item. The scores will therefore range from 7 to 49 for the negative scale..
  There are no cut-off points for the direct scores obtained, but these are transformed by means of a conversion table into percentiles. Futhermore, PANSS also provides categorical information, indicating whether the schizophrenic disorder is positive, negative or mixed.
Changes in Clinical Efficacy of Prebiotic/Probiotic Dietary Modulation in 6 Months of Intervention | Basal, three and six months respectively
  -- Scale for Positive and Negative Schizophrenia Syndrome (categorized PANSS): discrete. It provides four dimensional scores: Positive syndrome, Negative syndrome, Compound scale, General psychopathology.
  The score on the general psychopathology (PANSS-PG) scale is obtained by adding up the scores of each item. The scores will therefore rangd from 16 to 112 for the general psychopathology.
  There are no cut-off points for the direct scores obtained, but these are transformed by means of a conversion table into percentiles. Futhermore, PANSS also provides categorical information, indicating whether the schizophrenic disorder is positive, negative or mixed.
Changes in Clinical Efficacy of Prebiotic/Probiotic Dietary Modulation in 6 Months of Intervention | Basal, three and six months respectively
  -- Scale for Positive and Negative Schizophrenia Syndrome (categorized PANSS): discrete. It provides four dimensional scores: Positive syndrome, Negative syndrome, Compound scale, General psychopathology.
  The score on the composite scale (PANNS-C) is obtained by subtracting the score on the negative scale from the score on the positive scale. This scale can have positive or negative valence, ranging from -42 to + 42.
  There are no cut-off points for the direct scores obtained, but these are transformed by means of a conversion table into percentiles. Futhermore, PANSS also provides categorical information, indicating whether the schizophrenic disorder is positive, negative or mixed.
Changes in Adherence to the Proposed Dietary Pattern in 6 Months of Intervention | Basal and six months respectively
  -- Food Consumption Frequency Questionnaire (CFCA) result: continuous. For the proper analysis of this document, it is necessary to transform the answers obtained from the Food Consumption Frequency Questionnaire -FCA- into the number of times each item was consumed per week and into the number of times it was consumed per day. The g/day was then calculated by multiplying the frequencies of consumption of each item by the weight of the usual consumption ration of each item (Weight of Ration of Items table -PRI-). Finally, the energy and nutritional value was calculated by applying the Adapted Food Composition table (AFC): first the consumption in the population of all the foods included in each item was added; then, the proportion of this total provided by each of these foods was calculated
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Weight (kg, continuous).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Height (cm, continuous), circumference (cm, continuous).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - BMI: Weight and height will be combined to report BMI in kg/m^2 (continous).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Systolic blood pressure (mmHg, continuous), diastolic blood pressure (mmHg, continuous).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Heart rate (ppm, discrete).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Biochemical profile: glucose (mg/dL, discrete), cholesterol (mg/dL, discrete), triglycerides (mg/dL, discrete), C-HDL (mg/dL, discrete), C-LDL (mg/dL, discrete), total cholesterol/C-HDL (mg/dL, discrete).
Improvement on Cardiometabolic Profile | Every month, during 6 months of intervention
  - Biochemical profile: LDH (IU/L, discrete).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: Red blood cells (x10e6/mm3, continuous).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: Haemoglobin (g/dL, continuous), C.H.C.M. (g/dL, discrete).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: Haematocrit (%, continuous), R.D.W (%, continuous)..
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: M.C.V. (fL, discrete), M.P.V. (fL, discrete).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: H.C.M. (pg ,discrete).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: Leukocytes (x10e3/mm3, discrete).
Changes in Blood Test Variables in 6 Months of Intervention | Basal, three and six months respectively
  -- Haematological profile: Neutrophils (x10e3/m, continuous), lymphocytes (x10e3/m, continuous), monocytes (x10e3/m, continuous), eosinophils (x10e3/m, continuous), basophils (x10e3/m, continuous), platelets (x10e3/mm3, discrete).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile:
  ALT/GPT (IU/L, discrete), G-GT (IU/L, discrete), FAL (IU/L, discrete) a-HBs (UI/L, continuous), LUES (UI/L, nominal/discrete), a-HAV-M (UI/L, nominal/discrete), a-HCV (UI/L, nominal/discrete), HBsAg (UI/L, nominal/discrete), a-HBC-IgG (UI/L, nominal/discrete).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: Na+/K+ (mEq/L, discrete/continuous, respectively), Cl- (mEq/L, continuous), Ca2+ (mEq/L, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: Urate (mg/dL, continuous), creatinine (mg/dL, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: HbA1c (%, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: HbA1c IFCC (mmol/mol, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: Fructosamine (mcmol/L, discrete).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: Fe2+ (mcg/dL, discrete), FRT (mcg/dL, discrete), folate (mcg/dL, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile:Vit.B12 (ng/mL, discrete), vit.D total (D2+D3) 25-OH (ng/mL, discrete).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: Glomerular filtrate estimation (mL/min/1,73 m^2, discrete).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: TSH (mU/L, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile: PRL (ng/dL, continuous).
Changes in Other Biochemical Parameters | Basal, three and six months respectively
  - Biochemical profile:
  Na+/K+ (mEq/L, discrete/continuous, respectively), Cl- (mEq/L, continuous), Ca2+ (mEq/L, continuous),
Changes in Stool Culture in 6 Months of Intervention | Basal and six months respectively
  -- Stool Culture: General bacteriology - Usual mixed flora/disbiosis: Salmonella spp (nominal), Shigella spp (nominal), Yersinia spp (nominal), Hafnia alvei (nominal), Aermonas spp (nominal), Campylobacter spp (nominal) -.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Córdoba., Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
In the dissemination plan, it has been considered appropriate to share all the information on the protocol and questionnaires used in the development of the clinical trial.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Balanza Martinez V. Nutritional supplements in psychotic disorders. Actas Esp Psiquiatr. 2017 Sep;45(Supplement):16-25. Epub 2017 Sep 1. PMID 29171643
- [Background] American Psychiatric Association. Manual diagnóstico y estadístico de los trastornos mentales: DSM-5. Madrid: Editorial Médica Panamericana;2014.
- [Background] Gómez AE. Nutrición y enfermedad mental. Esquizofrenia y ácidos grasos omega 3. Farmacia Profesional. 2007;21(3):60-63
- [Background] Bernardo M, Canas F, Herrera B, Garcia Dorado M. Adherence predicts symptomatic and psychosocial remission in schizophrenia: Naturalistic study of patient integration in the community. Rev Psiquiatr Salud Ment. 2017 Jul-Sep;10(3):149-159. doi: 10.1016/j.rpsm.2016.04.001. Epub 2016 Jun 10. English, Spanish. PMID 27291833
- [Background] Tandon R, Nasrallah HA, Keshavan MS. Schizophrenia, "just the facts" 4. Clinical features and conceptualization. Schizophr Res. 2009 May;110(1-3):1-23. doi: 10.1016/j.schres.2009.03.005. Epub 2009 Mar 27. PMID 19328655
- [Background] Godoy JF, Caballero M, Godoy-Izquierdo D, Vázquez ML, Muela JA. Prevención de recaídas en la esquizofrenia: propuesta de un programa de intervención durante la fase prodrómica. Rei Do Crea. 2016;Vol.5(1):56-58. DOI 10.1016 / j.rcp.2015.05.011
- [Background] Soria V, Uribe J, Salvat-Pujol N, Palao D, Menchon JM, Labad J. Psychoneuroimmunology of mental disorders. Rev Psiquiatr Salud Ment (Engl Ed). 2018 Apr-Jun;11(2):115-124. doi: 10.1016/j.rpsm.2017.07.006. Epub 2017 Oct 6. English, Spanish. PMID 28993125
- [Background] Cepeda V, Mondragón A, Lamas A, Miranda JM, Cepeda A. Empleo de prebióticos y probióticos en el manejo de la ansiedad. Farmaceut Comunit. 2019;11(2):30-40. DOI:10.5672/FC.2173-9218
- [Background] Icaza-Chavez ME. [Gut microbiota in health and disease]. Rev Gastroenterol Mex. 2013 Oct-Dec;78(4):240-8. doi: 10.1016/j.rgmx.2013.04.004. Epub 2013 Nov 28. Spanish. PMID 24290319
- [Background] Castillo-Alvarez F, Marzo-Sola ME. Role of the gut microbiota in the development of various neurological diseases. Neurologia (Engl Ed). 2022 Jul-Aug;37(6):492-498. doi: 10.1016/j.nrl.2019.03.017. Epub 2019 Jul 21. English, Spanish. PMID 31340904
- [Background] Rodríguez A, Solano M. Nutrición y salud mental: revisión bibliográfica. Rev Post Psiquiat UNAH. 2008;1(3):1-5.
- [Background] Salagre E, Vieta E, Grande I. The visceral brain: Bipolar disorder and microbiota. Rev Psiquiatr Salud Ment. 2017 Apr-Jun;10(2):67-69. doi: 10.1016/j.rpsm.2017.02.001. Epub 2017 Mar 22. No abstract available. English, Spanish. PMID 28341435
- [Background] Wang HX, Wang YP. Gut Microbiota-brain Axis. Chin Med J (Engl). 2016 Oct 5;129(19):2373-80. doi: 10.4103/0366-6999.190667. PMID 27647198
- [Background] Mariño A, Núñez M, Barreto J. Microbiota, probióticos, prebióticos y simbióticos. Pediatr Integral. 2015; 19(5):337-354.
- [Background] Andreo P, García N, Sánchez EP. La microbiota intestinal y su relación con las enfermedades mentales a través del eje microbiota-intestino-cerebro. Rev Dis Cli Neuro. 2017;4(2):52-58.
- [Background] Kim YK, Shin C. The Microbiota-Gut-Brain Axis in Neuropsychiatric Disorders: Pathophysiological Mechanisms and Novel Treatments. Curr Neuropharmacol. 2018;16(5):559-573. doi: 10.2174/1570159X15666170915141036. PMID 28925886
- [Background] Patra S. Psychobiotics: A paradigm shift in psychopharmacology. Indian J Pharmacol. 2016 Jul-Aug;48(4):469-470. doi: 10.4103/0253-7613.186194. No abstract available. PMID 27756969
- [Background] Sarkar A, Lehto SM, Harty S, Dinan TG, Cryan JF, Burnet PWJ. Psychobiotics and the Manipulation of Bacteria-Gut-Brain Signals. Trends Neurosci. 2016 Nov;39(11):763-781. doi: 10.1016/j.tins.2016.09.002. Epub 2016 Oct 25. PMID 27793434
- [Background] Kali A. Psychobiotics: An emerging probiotic in psychiatric practice. Biomed J. 2016 Jun;39(3):223-4. doi: 10.1016/j.bj.2015.11.004. Epub 2016 Aug 9. PMID 27621125
- [Background] Forsythe P, Kunze W, Bienenstock J. Moody microbes or fecal phrenology: what do we know about the microbiota-gut-brain axis? BMC Med. 2016 Apr 19;14:58. doi: 10.1186/s12916-016-0604-8. PMID 27090095
- [Background] Galletero JM. Nutrición y enfermedad mental. Marcadores bioquímicos en el trastorno bipolar. Zainak. 2011;34:323-334
- [Background] Franch CM, Molina V, Franch JI. Factores determinantes del riesgo metabólico en el tratamiento con antipsicóticos atípicos. Rev Psiquiatr Salud Ment. 2016;23(3):87-130. DOI: 10.1016/j.psiq.2016.08.001
- [Background] Franch Pato CM, Molina Rodriguez V, Franch Valverde JI. Metabolic syndrome and atypical antipsychotics: Possibility of prediction and control. Rev Psiquiatr Salud Ment. 2017 Jan-Mar;10(1):38-44. doi: 10.1016/j.rpsm.2016.09.003. Epub 2016 Dec 7. English, Spanish. PMID 27939025
- [Background] Sánchez ML, González J, Martínez MC. Control metabólico y prolactina en la enfermedad mental grave. Intervenciones enfermeras. Rev Enferm Salud Ment. 2018;9:24-28. DOI: 10.5538/2385-703X.2018.9.24
- [Background] Pringsheim T, Kelly M, Urness D, Teehan M, Ismail Z, Gardner D. Physical Health and Drug Safety in Individuals with Schizophrenia. Can J Psychiatry. 2017 Sep;62(9):673-683. doi: 10.1177/0706743717719898. Epub 2017 Jul 18. PMID 28718324
- [Background] Pina-Camacho L, Diaz-Caneja CM, Saiz PA, Bobes J, Corripio I, Grasa E, Rodriguez-Jimenez R, Fernandez M, Sanjuan J, Garcia-Lopez A, Tapia-Casellas C, Alvarez-Blazquez M, Fraguas D, Mitjans M, Arias B, Arango C. Pharmacogenetic study of second-generation antipsychotic long-term treatment metabolic side effects (the SLiM Study): rationale, objectives, design and sample description. Rev Psiquiatr Salud Ment. 2014 Oct-Dec;7(4):166-78. doi: 10.1016/j.rpsm.2014.05.004. Epub 2014 Oct 19. English, Spanish. PMID 25440735
- [Background] Severi E, Ferrara M, Tedeschini E, Vacca F, Mungai F, Amendolara R, Baccari F, Starace F. Assessment of cardiovascular risk in an Italian psychiatric outpatient sample: A chart review of patients treated with second-generation antipsychotics. Int J Ment Health Nurs. 2018 Jun;27(3):1002-1008. doi: 10.1111/inm.12407. Epub 2017 Dec 2. PMID 29197134
- [Background] Ocando L, Roa A, León M, González R. Antipsicóticos atípicos y su papel en el desarrollo de enfermedades metabólicas. Rev Iberoam Hipert. 2018;13(2):44-51.
- [Background] Gurusamy J, Gandhi S, Damodharan D, Ganesan V, Palaniappan M. Exercise, diet and educational interventions for metabolic syndrome in persons with schizophrenia: A systematic review. Asian J Psychiatr. 2018 Aug;36:73-85. doi: 10.1016/j.ajp.2018.06.018. Epub 2018 Jun 30. PMID 29990631
- [Background] Cortés B. Síndrome metabólico y antipsicóticos de segunda generación. Rev Asoc Esp Neuropsiq. 2011;31(110):303-320. DOI: 10.4321/S0211-57352011000200009
- [Background] Gonzalez Jimenez E. Obesity: etiologic and pathophysiological analysis. Endocrinol Nutr. 2013 Jan;60(1):17-24. doi: 10.1016/j.endonu.2012.03.006. Epub 2012 May 22. English, Spanish. PMID 22622157
- [Background] Chee GL, Wynaden D, Heslop K. Improving metabolic monitoring rate for young people aged 35 and younger taking antipsychotic medications to treat a psychosis: A literature review. Arch Psychiatr Nurs. 2017 Dec;31(6):624-633. doi: 10.1016/j.apnu.2017.09.002. Epub 2017 Sep 6. PMID 29179831
- [Background] Sanchez-Martinez V, Romero-Rubio D, Abad-Perez MJ, Descalzo-Cabades MA, Alonso-Gutierrez S, Salazar-Fraile J, Montagud V, Facila L. Metabolic Syndrome and Cardiovascular Risk in People Treated with Long-Acting Injectable Antipsychotics. Endocr Metab Immune Disord Drug Targets. 2018;18(4):379-387. doi: 10.2174/1871530317666171120151201. PMID 29165095
- [Background] Pérez BY, Jasso JA, López MM. Evaluación del estado nutricio en pacientes con trastornos psiquiátricos en una unidad hospitalaria. Nutr Clín Diet Hosp. 2017; 37(1):24-33. DOI: 10.12873/371brendayadira
- [Background] Consejería de Salud. Consejo Dietético en Atención Primaria. Plan para la Promoción de la Salud Física y la Alimentación Equilibrada 2004-2008. Consejería de Salud. Junta de Andalucía; 2010. [Internet]. 2010. [access 6 november 2019]. Available from: https://www.juntadeandalucia.es/organismos/saludyfamilias/areas/saludvida/adulta/paginas/conscon-dietetico.html
- [Background] Consejería de Salud. Guía de Consejo Dietético Intensivo en Atención Primaria. Plan para la Promoción de la Salud Física y la Alimentación Equilibrada 2004-2008. Consejería de Salud. Junta de Andalucía; 2007. [Internet]. 2007. [access 10 november 2019]. Available from: https://www.juntadeandalucia.es/organismos/saludyfamilias/areas/saludvida/adulta/paginas/consejo-dietetico.html
- [Background] Agencia Española de Seguridad Alimentaria y Nutrición (AESAN) [sede Web]. Madrid: AECOSAN; 2015- [updated 12 november 2019; access el 14 november 2019]. Available from: http://www.aecosan.msssi.gob.es/AECOSAN/web/home/aecosan_inicio.htm
- [Background] Hamui A, Varela M. La técnica de grupos focales. Inv Ed Med. 2013; 2(1):55-60. DOI: 10.1016/S2007-5057(13)72683-8
- [Background] Martin-Moreno JM, Boyle P, Gorgojo L, Maisonneuve P, Fernandez-Rodriguez JC, Salvini S, Willett WC. Development and validation of a food frequency questionnaire in Spain. Int J Epidemiol. 1993 Jun;22(3):512-9. doi: 10.1093/ije/22.3.512. PMID 8359969
- [Background] Junta de Andalucía. Instrumento de evaluación nº 8: Detección e intervención temprana en las psicosis. Escala para el síndrome positivo y negativo de la esquizofrenia (PANSS). Servicio Andaluz de Salud; 2010. [Internet]. 2010. [access 5 november 2019]. Available from: http://http://www.sspa.juntadeandalucia.es/servicioandaluzdesalud/publicaciones/listadodetalle.asp?idp=433
- [Background] Garcia-Portilla MP, Saiz PA, Bousono M, Bascaran MT, Guzman-Quilo C, Bobes J; en nombre del grupo de validacion de la version espanola de la escala de Funcionamiento Personal y Social (PSP). Validation of the Spanish Personal and Social Performance scale (PSP) in outpatients with stable and unstable schizophrenia. Rev Psiquiatr Salud Ment. 2011 Jan;4(1):9-18. doi: 10.1016/j.rpsm.2010.11.003. Epub 2011 Mar 10. English, Spanish. PMID 23446097
- [Background] Sugawara N, Sagae T, Yasui-Furukori N, Yamazaki M, Shimoda K, Mori T, Sugai T, Matsuda H, Suzuki Y, Ozeki Y, Okamoto K, Someya T. Effects of nutritional education on weight change and metabolic abnormalities among patients with schizophrenia in Japan: A randomized controlled trial. J Psychiatr Res. 2018 Feb;97:77-83. doi: 10.1016/j.jpsychires.2017.12.002. Epub 2017 Dec 5. PMID 29220825
- [Background] Carmenate L, Moncada FE, Borjas WE. Manual de medidas antropométricas. 1ª ed. Costa Rica: SALTRA, 2014.
- [Derived] Sevillano-Jimenez A, Romero-Saldana M, Garcia-Mellado JA, Carrascal-Laso L, Garcia-Rodriguez M, Molina-Luque R, Molina-Recio G. Impact of high prebiotic and probiotic dietary education in the SARS-CoV-2 era: improved cardio-metabolic profile in schizophrenia spectrum disorders. BMC Psychiatry. 2022 Dec 12;22(1):781. doi: 10.1186/s12888-022-04426-9. PMID 36510155
- [Derived] Sevillano-Jimenez A, Molina-Recio G, Garcia-Mellado JA, Garcia-Rodriguez M, Molina-Luque R, Romero-Saldana M. Efficacy of nutrition education for the increase of symbiotic intake on nutritional and metabolic status in schizophrenic spectrum disorders: A two-arm protocol. Front Nutr. 2022 Aug 10;9:912783. doi: 10.3389/fnut.2022.912783. eCollection 2022. PMID 36034912
- See also: Junta de Andalucía. Instrumento de evaluación nº 8: Detección e intervención temprana en las psicosis. Escala para el síndrome positivo y negativo de la esquizofrenia (PANSS). Servicio Andaluz de Salud — http://www.sspa.juntadeandalucia.es/servicioandaluzdesalud/publicaciones/listadodetalle.asp?idp=433